CLINICAL TRIAL: NCT00709423
Title: A Randomized, Double-Masked, Placebo-Controlled Two Cross Over Study Comparing the Effects of Moxaverine and Placebo on Ocular Blood Flow
Brief Title: Effects of Moxaverine and Placebo on Ocular Blood Flow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dorothea Gross, Ursapharm, Germany
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPHT-161106
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-06

CONDITIONS: Regional Blood Flow; Ocular Physiology; Retina
MeSH Terms: interventions — moxaverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Moxaverine; Drug: Moxaverin 150mg
- 2 (Placebo Comparator)
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: Moxaverine
  Arms: 1
Drug: Moxaverin 150mg — intravenous administration
  Other Names: Collateral i
  Arms: 1
Drug: NaCl — intravenous administration
  Arms: 2

SUMMARY:
A number of common eye diseases such as retinal artery and vein occlusion, diabetic retinopathy, age-related macular degeneration, glaucoma and anterior ischemic optic neuropathy are associated with ocular perfusion abnormalities. Although this is well recognized there is not much possibility to improve blood flow to the posterior pole of the eye in these diseases.

Since many years, moxaverine is used in the therapy of perfusion abnormalities in the brain, the heart and the extremities. This is based on a direct vasodilator effect of the drug, but also on the rheological properties of red blood cells. Whether moxaverine affects blood flow in the eye is unknown. The present study aims to investigate whether moxaverine may improves blood flow in the eye after systemic administration.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages or drugs, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Ametropy >= 3 dpt
* Acute gastric bleeding, massive cerebral hemorrhage related to stroke
* Women: pregnancy or lactation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Retinal blood flow (Laser Doppler Velocimetry, Retinal Vessel Analyzer) | 2 hours
Choroidal and optic nerve head blood flow (Laser Doppler Flowmetry) | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clincal Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clincal Pharmacology, Medical University of Vienna, Vienna, Austria